CLINICAL TRIAL: NCT02376608
Title: Pronovum - An Open-label, Randomized, Single-dose Study to Evaluate the Bioavailability of Omega-3 Food Supplements in Healthy Male and Female Subjects.
Brief Title: Bioavailability of Omega-3 Food Supplement in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pronova BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CTN00714101
Record Dates: First submitted 2015-02-10; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2014-08

CONDITIONS: Biological Availability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pronova Pure 150:500 EE EU (Active Comparator): 2 × PronovaPure 150:500 EE EU
  Interventions: Dietary Supplement: Pronova Pure 150:500 EE EU; Dietary Supplement: Pronovum PRF-037; Dietary Supplement: Pronovum PRF-041; Dietary Supplement: Eskimo-3
- Pronovum PRF-037 (Active Comparator): 2 × Pronovum PRF-037
  Interventions: Dietary Supplement: Pronova Pure 150:500 EE EU; Dietary Supplement: Pronovum PRF-037; Dietary Supplement: Pronovum PRF-041; Dietary Supplement: Eskimo-3
- Pronovum PRF-041 (Active Comparator): 2 × Pronovum PRF-041
  Interventions: Dietary Supplement: Pronova Pure 150:500 EE EU; Dietary Supplement: Pronovum PRF-037; Dietary Supplement: Pronovum PRF-041; Dietary Supplement: Eskimo-3
- Eskimo-3 (Active Comparator): 3 × Eskimo-3
  Interventions: Dietary Supplement: Pronova Pure 150:500 EE EU; Dietary Supplement: Pronovum PRF-037; Dietary Supplement: Pronovum PRF-041; Dietary Supplement: Eskimo-3

INTERVENTIONS:
Dietary Supplement: Pronova Pure 150:500 EE EU — Each subject will participate in 4 treatment periods. The subjects are randomized to one of the following treatment sequences ABCD, BDAC, CADB, DCBA. 4 treatment free days between each treatment period
Dietary Supplement: Pronovum PRF-037 — Each subject will participate in 4 treatment periods. The subjects are randomized to one of the following treatment sequences ABCD, BDAC, CADB, DCBA. 4 treatment free days between each treatment period
Dietary Supplement: Pronovum PRF-041 — Each subject will participate in 4 treatment periods. The subjects are randomized to one of the following treatment sequences ABCD, BDAC, CADB, DCBA. 4 treatment free days between each treatment period
Dietary Supplement: Eskimo-3 — Each subject will participate in 4 treatment periods. The subjects are randomized to one of the following treatment sequences ABCD, BDAC, CADB, DCBA. 4 treatment free days between each treatment period

SUMMARY:
The study will evaluate the relative bioavailability of Pronovum PRF-037 and Pronovum PRF-041 with PronovaPure 150:150 EE EU and Eskimo-3 (500 mg omega-3 acid triglyceride containing 80 mg EPA and 50 mg DHA per gram oil) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* males or females
* any ethnic origin
* BMI 18.5 - 30.0 kg/m2
* generally in good health
* signed informed consent

Exclusion Criteria:

* males or females not willing to use appropriate contraception
* prescribed systemic or topical medication within 14 days and slow release medication considered to be active within 14 days.
* omega-3 fatty acids or fish oil within 2 weeks of dosing.
* any non-prescribed systemic or topical medication including herbal remedies and vitamin/mineral supplements within 7 days
* any medication incl. St.John's Worth known to chronically alter drug absorption/elimination within 30 days
* Subjects still present in clinical study or in the past 3 months
* recent blood donation
* drug allergy or significant allergic disease
* allergic or hypersensitivity to omega-3 acids, fish, soya, oleic acid, sesame oil or other constituents in pharma preparation
* high consumption of alcohol
* high consumption of tobacco
* hepatitis or HIV
* vegetarians
* earlier participated in or withdrawn from the study
* not willing to follow dietary restrictions
* frequent occurence of migraine attacks
* subjects that should not participate according to investigator

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Area under curve of omega-3 food supplements under light fed conditions in healthy subjects. | Pharmacikinetics up to 36 hours post-dose
Peak plasma concentration of omega-3 food supplements under light fed conditions in healthy subjects. | Pharmacikinetics up to 36 hours post-dose

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability. | During entire study period, an expected average of 7 weeks from screening to last visit.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Strong, MD, Principal Investigator — Covance Clinical Research Unit (CRU) Ltd.
Locations (1):
- Covance Clinical research Unit (CRU) Ltd,Springfield House, Hyde street, Leeds, United Kingdom